CLINICAL TRIAL: NCT06372691
Title: How Do We Ultrasound-Guided Popliteal Approach Sciatic Nerve Block;Is It Injection Subparaneural, Interneural?
Brief Title: How Do We Ultrasound-Guided Popliteal Approach Sciatic Nerve Block?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, semih başkan, Doç. Prof. Dr., Ankara City Hospital Bilkent
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: PoplitealApproach SciaticBlock
Record Dates: First submitted 2024-04-01; First posted 2024-04-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2024-09

CONDITIONS: Adult; Regional Anesthesia Morbidity; Anesthesia Injection Site
Keywords: Popliteal Approach Sciatic Nerve Block; Regional Anesthesia; Foot, Ankle and Toe Amputation
MeSH Terms: interventions — Dental Occlusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Subparaneural Injection (Group S) (Active Comparator): The position of the patients will be prone.The skin will be cleaned according to asepsis and antisepsis rules.After preparing the USG a high-frequency linear array transducer under sterile conditions,we will be positioned it transversely in the popliteal fossa.After visualizing the artery,its hyperechoic nerves will be founded superficially.The sciatic nerve will be identified proximally to visualize where the TN and CPN eventually come together to form the sciatic nerve and separate distally where the CPN moves laterally and the TN remains medially.Once the nerves began to separate,they will be scanned until a figure 8 or pant leg image will be obtained.Using the in-plane technique under ultrasonography guidance, injection will be applied to the subparaneural area in Group S.1 ml of LA solution was injected for the purpose of verifying proper needle insertion.A standard dose of 15 mL bupivacaine 0.5% and 5mg/mL local anesthetic was used accompanied by a 20G,12mm block needle.
  Interventions: Other: Subparaneural Injection (Grup S), Block
- Interneural Injection (Group I) (Active Comparator): The position of the patients will be prone.The skin will be cleaned according to asepsis and antisepsis rules.After preparing the USG a high-frequency linear array transducer under sterile conditions, we will be positioned it transversely in the popliteal fossa.After visualizing the artery, its hyperechoic nerves will be founded superficially.The sciatic nerve will be identified proximally to visualize where the TN and CPN eventually come together to form the sciatic nerve and separate distally where the CPN moves laterally and the TN remains medially.Once the nerves began to separate, they will be scanned until a figure 8 or pant leg image will be obtained.Using the in-plane technique under ultrasonography guidance, injection will be applied to the interneural area in Group I.1 ml of LA solution was injected for the purpose of verifying proper needle insertion.A standard dose of 15 mL bupivacaine 0.5% and 5mg/mL local anesthetic was used accompanied by a 20 G, 12mm block needle.
  Interventions: Other: Interneural Injection (Grup I), Block

INTERVENTIONS:
Other: Subparaneural Injection (Grup S), Block — Comparison of two different methods in terms of various features
  Arms: Subparaneural Injection (Group S)
Other: Interneural Injection (Grup I), Block — Comparison of two different methods in terms of various features
  Arms: Interneural Injection (Group I)

SUMMARY:
The aim of this prospective, randomized, observer-blind study to compare subparaneural approach injection with interneural approach injection in popliteal sciatic nerve blocks.

DETAILED DESCRIPTION:
The study will involve American Society of Anesthesiologists Physical Status Classification (ASA) III or IV risk group patients, 18 years of age or older, who will undergoing foot, ankle, or toe amputation.

Supparaneural injection (Group S) and interneural injection method (Group I) will the two research groups to which patients were randomly allocated.

Every 5 minutes following LA injection, an investigator who will blind to randomization will assess the sensory and motor blockage in the operated foot. The study will documented the operative time, block characteristics, such as the duration of block administration, sensory and motor block start and regression times, the time of extra analgesic required, and the occurrence of complications.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and over
* Planned foot, ankle or toe amputation
* ASA III-IV risk group
* Patients who agreed to be included in the study

Exclusion Criteria:

* People with neurological and psychiatric diseases
* Using opioids or another analgesic for chronic pain
* Allergic to local anesthetics
* Pregnant or breastfeeding
* Those with infection or sepsis in the application area
* Patients who did not agree to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Onset Time | Time from the moment the block is made to the moment it starts, within the first half hour
  Onset time will be defined as the moment when it is determined that the block is successful.

SECONDARY OUTCOMES:
Block Execution Times | 1-10 minutes
  The time from the moment the block starts to the moment the transaction ends.
Need for Multiple Injections Owing to Insufficient Anesthesia | Within 24 hours
  How many blocks should be made.
Additional Rescue Analgesic | Within 24 hours
  Analgesic use status.
Adverse Effects to Anesthesia | During the block period, within 24 hours
  hypotension, agitation, nausea, vomiting, dizziness
Hemodynamic Effects Of The Block | 0th minutes, 5th minutes,10th minutes,15th minutes,20th minutes,25th minutes,30th minutes,35th minutes,40th minutes,45th minutes,50th minutes,55th minutes and 60th minutes and then at 1-hour intervals and 15th minutes,30th minutes
  Noninvasive systolic and diastolic blood pressure
Effects Of The Block On Heart Rate | 0th minutes, 5th minutes,10th minutes,15th minutes,20th minutes,25th minutes,30th minutes,35th minutes,40th minutes,45th minutes,50th minutes,55th minutes and 60th minutes and then at 1-hour intervals and 15th minutes,30th minutes
  Heart rate
Effects Of The Block On Peripheral Pulse Oximetry | 0th minutes, 5th minutes,10th minutes,15th minutes,20th minutes,25th minutes,30th minutes,35th minutes,40th minutes,45th minutes,50th minutes,55th minutes and 60th minutes and then at 1-hour intervals and 15th minutes,30th minutes
  Peripheral pulse oximetry
Regression Time Of Sensory and Motor Block | Within 24 hours
  When the block starts to come back.
Total Block Times | Within 24 hours
  How long the block took in total.

CONTACTS AND LOCATIONS:
Overall Officials: Semih Başkan, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital, Ankara, Çankaya, Turkey (Türkiye)